CLINICAL TRIAL: NCT05977959
Title: Optimizing the Impact of the Healthy School Recognized Campus Program on Youth's CVD Risk Factors
Acronym: HSRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AHA HSRC
Record Dates: First submitted 2023-07-24; First posted 2023-08-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Physical Activity; Nutrition
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Mentoring Program (Experimental): Participants in this group will receive the Mentoring Program strategy in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Mentoring Program
- Enhanced Resources (Experimental): Participants in this group will receive the Enhanced Resources strategy in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Enhanced Resources
- Enhanced Engagement (Experimental): Participants in this group will receive the Enhanced Engagement strategy in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Enhanced Engagement
- No Intervention (No Intervention): All schools will participate in the HSRC initiative. The requirements for the initiative are to complete a school-wide walking program, 1 youth, and 1 adult program from a list of available programs that make up the initiative.
- Mentoring + Enhanced Resources (Experimental): Participants in this group will receive the Mentoring Program and Enhanced Resources strategies in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Mentoring Program; Behavioral: Enhanced Resources
- Mentoring + Enhanced Engagement (Experimental): Participants in this group will receive the Mentoring Program and Enhanced Engagement strategies in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Mentoring Program; Behavioral: Enhanced Engagement
- Enhanced Resources + Enhanced Engagement (Experimental): Participants in this group will receive the Enhanced Resources and Enhanced Engagement strategies in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Enhanced Resources; Behavioral: Enhanced Engagement
- Mentoring + Enhanced Resources + Enhanced Engagement (Experimental): Participants in this group will receive the Mentoring Program, Enhanced Resources, and Enhanced Engagement strategies in addition to Healthy School Recognized Campus.
  Interventions: Behavioral: Mentoring Program; Behavioral: Enhanced Resources; Behavioral: Enhanced Engagement

INTERVENTIONS:
Behavioral: Mentoring Program — Schools in this group will participate in meetings and discussion boards and receive newsletters to help with program implementation.
  Arms: Mentoring + Enhanced Engagement; Mentoring + Enhanced Resources; Mentoring + Enhanced Resources + Enhanced Engagement; Mentoring Program
Behavioral: Enhanced Resources — Schools in this group will receive extra resources such as program incentives to aid in program implementation.
  Arms: Enhanced Resources; Enhanced Resources + Enhanced Engagement; Mentoring + Enhanced Resources; Mentoring + Enhanced Resources + Enhanced Engagement
Behavioral: Enhanced Engagement — Schools in this group will participate in program contests to aid program implementation.
  Arms: Enhanced Engagement; Enhanced Resources + Enhanced Engagement; Mentoring + Enhanced Engagement; Mentoring + Enhanced Resources + Enhanced Engagement

SUMMARY:
Healthy School Recognized Campus is a Texas A&M AgriLife Extension initiative that supports the delivery of school-based physical activity and nutrition programs for diverse youth across Texas. The purpose of this study is to improve the delivery of these programs and optimize the effect they have on youth's cardiovascular risk factors.

DETAILED DESCRIPTION:
The investigators will conduct a group randomized factorial trial using the Multiphase Optimization STrategy (MOST) framework to evaluate the impact (i.e., implementation and effectiveness) of three implementation strategies on program implementation and youth's cardiovascular disease risk. HSRC is a Texas A&M AgriLife Extension initiative that supports the delivery of school-based physical activity and nutrition programs.

Elementary schools in North and East Texas (n=16) of similar socio-economic status will be randomized at baseline to receive either 3, 2, 1, or no strategies to support HSRC program implementation. All schools will participate in HSRC during the full school year.

The investigators hypothesize that one strategy will result in significantly greater HSRC implementation and effectiveness than the other strategies tested.

ELIGIBILITY:
School Inclusion Criteria:

* located in North and East Texas
* Public elementary school

Student Inclusion Criteria"

* at least 10 years old by September 1, 2023 (2024 for the 2024-2025 school year)
* enrolled in the 5th or 6th grade
* able to read, speak, and write in English

Exclusion Criteria:

* any motor or cognitive impairments or other health conditions that would prevent them from completing a physical assessment

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Presence or absence of metabolic syndrome (MetS) | Baseline, 9 months (immediate post intervention)
  MetS is present after identifying abdominal obesity plus at least two of the four other MetS Risk factors: high blood pressure, high blood sugar, low HDL cholesterol, and high triglyceride levels.
  MetS = (abdominal obesity) + (2 of 4 other MetS Risk factors)
  Measures to determine MetS risk factors:
  1. Abdominal obesity: waist circumference >90th percentile for child's sex and age
  2. High blood pressure: systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥90 mmHg)
  3. High blood glucose: blood glucose ≥5.6 mmol/L or known diabetes
  4. Low HDL cholesterol: HDL cholesterol <1.03 mmol/L
  5. High triglyceride level: Triglyceride level ≥ 1.7mmol/L
Change in the number of MetS risk factors | Baseline, 9 months (immediate post intervention)
  Change in the number of MetS risk factors = (new # of MetS risk factors) - (original # of MetS risk factors)
  Measures to determine MetS risk factors:
  1. Abdominal obesity: waist circumference >90th percentile for child's sex and age
  2. High blood pressure: systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥90 mmHg)
  3. High blood glucose: blood glucose ≥5.6 mmol/L or known diabetes
  4. Low HDL cholesterol: HDL cholesterol <1.03 mmol/L
  5. High triglyceride level: Triglyceride level ≥ 1.7mmol/L
Number of programs schools delivered (in addition to Walk Across Texas) | Baseline, 9 months (immediate post intervention)
Number of sessions delivered for each program | Baseline, 9 months (immediate post intervention)
Length of the sessions delivered | Baseline, 9 months (immediate post intervention)
Individual-level attendance data for programs delivered | Baseline, 9 months (immediate post intervention)
Body mass index (BMI) | Baseline, 9 months (immediate post intervention)
  Weight will be measured with a scale (in pounds), and height will be measured using a stadiometer (in inches). Weight and height will be combined to report BMI as follows, BMI = (weight (lb)/height (inches)2) x 703.
Concentration of subdermal carotenoids | Baseline, 9 months (immediate post intervention)
  The concentration of subdermal carotenoids will assess the changes in fruit and vegetable consumption using the Veggie Meter: A non-invasive, portable machine that measures subdermal carotenoid levels using resonance Raman spectroscopy.
Physical fitness capacity estimation | Baseline, 9 months (immediate post intervention)
  Physical fitness will be measured using the FitnessGram PACER multistage aerobic capacity test: Children will run back and forth 20 meters, with an initial running speed of 8.5 km/hour and a progressive 0.5-km/hour increase in running speed every minute. As the test continues it becomes progressively harder. The number of laps completed is used to estimate children's physical fitness physical fitness.

SECONDARY OUTCOMES:
Blood pressure level | Baseline, 9 months (immediate post intervention)
  Blood pressure (systolic and diastolic) will be measured with two numbers using an automated Omron sphygmomanometer.
Concentration of blood glucose | Baseline, 9 months (immediate post intervention)
  Glucose will be measured using a portable CardioChek Plus analyzer to assess a single capillary blood sample following an overnight fast.
Waist circumference | Baseline, 9 months (immediate post intervention)
  Waist circumference will be measured at the midpoint between the floating rib and iliac crest using a tape measure.
Concentration of HDL cholesterol | Baseline, 9 months (immediate post intervention)
  HDL-C will be measured using a portable CardioChek Plus analyzer to assess a single capillary blood sample following an overnight fast.
Concentration of serum triglycerides | Baseline, 9 months (immediate post intervention)
  Triglycerides will be measured using a portable CardioChek Plus analyzer to assess a single capillary blood sample following an overnight fast.
Height | Baseline, 9 months (immediate post intervention)
  Height will be measured using a stadiometer in inches.
Weight | Baseline, 9 months (immediate post intervention)
  Weight will be measured with a scale in pounds.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Szeszulski, PhD, Principal Investigator — Texas A&M AgriLife
Locations (1):
- Texas A&M AgriLife Dallas Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Szeszulski J, Schaefers A, De Mello GT, Gardner J, George A, MacMillan Uribe A, Rethorst CD, Seguin-Fowler RA, Xin L. Design and methodology of a cluster randomized factorial trial to optimize implementation strategies for the Healthy School Recognized Campus initiative. Front Public Health. 2025 Oct 30;13:1652485. doi: 10.3389/fpubh.2025.1652485. eCollection 2025. PMID 41246086